CLINICAL TRIAL: NCT02100579
Title: Ultrasound-guided Adductor Canal Block for Total Knee Replacement: a Randomized, Double-blind Placebo Controlled Trial.
Brief Title: Ultrasound-guided Adductor Canal Block for Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Antoun Nader, Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00088239; STU00088239 (Other: Northwestern University IRB)
Record Dates: First submitted 2014-03-25; First posted 2014-04-01 (Estimated); Results first posted 2016-11-02 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Complications; Arthroplasty; Knee Injuries
MeSH Terms: conditions — Knee Injuries | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Group (Active Comparator): Ultrasound-guided adductor canal blockade with 10 ml of 0.25% bupivacaine
  Interventions: Drug: Bupivacaine
- Control Group (Placebo Comparator): Ultrasound-guided sham block with 10 ml of preservative free normal saline
  Interventions: Drug: Preservative free normal saline

INTERVENTIONS:
Drug: Bupivacaine — 10 ml of 0.25% bupivacaine
  Other Names: Sensorcaine
  Arms: Active Group
Drug: Preservative free normal saline — 10 ml of preservative free normal saline
  Other Names: 0.9% sodium chloride
  Arms: Control Group

SUMMARY:
Total knee arthroplasty is associated with intense early postoperative pain. Fast track recovery programs including early therapy protocols and early hospital discharge are being implemented at various hospitals. The postoperative analgesic pain regimen should enhance functional recovery in addition to providing efficient analgesia with minimal side effects. Adductor canal blockade is commonly used to provide postoperative analgesia for total knee arthroplasty (TKA) surgery. The investigators hypothesize that an ultrasound guided adductor canal block will lower narcotic consumption and improved overall satisfaction compared to ultrasound guided sham block with normal saline (placebo) for patients undergoing minimally invasive TKA surgery.

DETAILED DESCRIPTION:
The investigators hypothesize that an ultrasound guided adductor canal block will lower narcotic consumption and improved overall satisfaction compared to ultrasound guided sham block with normal saline (placebo) for patients undergoing minimally invasive TKA surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants 40 to 75 years old who are presenting for minimally invasive total knee arthroplasty under spinal anesthesia

Exclusion Criteria:

* Patient refusal
* American Society of Anesthesiologists physical status classification of 4 or higher
* Pre-existing neuropathy in the femoral or sciatic distribution
* Coagulopathy
* Infection at the site
* Chronic opioid use (greater than 3 months)
* Pregnancy
* Medical conditions limiting physical therapy participation
* Any other contra-indication to regional anesthesia

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoun Nader, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Group | Control Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Group | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 12 | 11 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [62 to 73] | 67 [59 to 72] | 67 [62 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption (mg morEq)
Description: Opioid consumption (morphine equivalents)
Time Frame: 36 hours
Measure: Median (Inter-Quartile Range); unit: Morphine Equivalents
Arm/Group | Active Group | Control Group
Number analyzed (Participants) | 20 | 20
Morphine Equivalents | 48 [39 to 61] | 60 [49 to 85]

2. Secondary Outcome: Visual Analog Scale Pain Score
Description: Visual Analog Scale pain score; 0 = no pain, 10 = excruciating pain) in the knee recorded every 6 hours up to 36hrs following surgery.
Time Frame: Pain burden at 36hr
Measure: Median (Inter-Quartile Range); unit: scores*hours
Arm/Group | Active Group | Control Group
Number analyzed (Participants) | 20 | 20
scores*hours | 71 [37 to 120] | 131 [92 to 161]

3. Secondary Outcome: Length of Hospitalization
Description: The average time to discharge in hours. Participants were discharged home went physical therapy criteria were met.
Time Frame: 0 to 192 hours
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Active Group | Control Group
Number analyzed (Participants) | 20 | 20
hours | 73 [64 to 83] | 92 [76 to 111]

ADVERSE EVENTS:
Arm/Group | Active Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes